CLINICAL TRIAL: NCT03991585
Title: Feasibility of the Musical Contour Regulation Facilitation (MCRF) Intervention to Promote Emotion Regulation in At-risk Preschoolers: A Clinical Pilot Study
Brief Title: MCRF Clinical Pilot Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: American Music Therapy Association (Other); University of Kansas (Other)
Responsible Party: Principal Investigator, Kimberly Sena Moore, Assistant Professor of Professional Practice, University of Miami
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 20190108
Record Dates: First submitted 2019-06-17; First posted 2019-06-19 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Emotional Adjustment
Keywords: At-risk preschoolers; Head Start; Emotion regulation
MeSH Terms: conditions — Emotional Regulation

STUDY DESIGN:
Intervention Model Description: There are six classroom assignments. Classrooms will be randomized to either of the treatment arms.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Three times a week MCRF (Experimental): Participants in this arm will participate in the MCRF intervention sessions three times a week for 12 consecutive weeks.
  Interventions: Behavioral: Musical Contour Regulation Facilitation (MCRF)
- One time a week MCRF (Experimental): Participants in this arm will participate in the MCRF intervention sessions one time a week for 12 consecutive weeks.
  Interventions: Behavioral: Musical Contour Regulation Facilitation (MCRF)

INTERVENTIONS:
Behavioral: Musical Contour Regulation Facilitation (MCRF) — MCRF involves 20-minute music therapy sessions comprised of seven interconnected components. Each session follows the same contour of neutral, low, and high arousal experiences facilitated through music.

SUMMARY:
The purpose of this study is to see if music can help children practice how to manage their emotions.

ELIGIBILITY:
Inclusion Criteria:

* Preschoolers aged 3 to 5 years old enrolled in a Head Start program
* Must be able to speak fluent English
* Must not have previously received music therapy services
* Must regularly attend the Head Start program
* Must have signed parental consent.

Exclusion Criteria:

* Does not meet all inclusion criteria

Ages: 3 Years to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 44 (Actual)
Dates: Start 2019-07-24 (Actual); Primary Completion 2020-01-15 (Actual); Study Completion 2020-01-15 (Actual)

PRIMARY OUTCOMES:
Change in emotion regulation as measured by Emotion Regulation Checklist (ERC) | Baseline, 12 weeks
  The Emotion Regulation subscale of the ERC is an 8-item, four-point Likert-type scale to assess ER processes in children. Parents and teachers will complete the ERC pre- and post-intervention. Scores range from 8 to 32 points. Higher scores reflect greater emotion regulation.
Change in emotional lability/negativity as measured by Emotion Regulation Checklist (ERC) | Baseline, 12 weeks
  The Lability/Negativity subscale of the ERC is a 15-item, four-point Likert-type scale to assess emotional lability in children. Parents and teachers will complete the ERC pre- and post-intervention. Scores range from 15 to 60 points. Higher scores reflect greater emotional lability.
Change in behaviors as measured by the Child Behavior Checklist for Ages 1.5-5 (CBCL/1.5-5) | Baseline, 12 weeks
  The CBCL/1.5-5 is a 99-item, three-point Likert-type scale to assess internalizing behaviors, externalizing behaviors, attending behaviors, and aggressive in preschool-aged children. Parents will complete the CBCL/1.5-5 pre- and post-intervention. Scores range from 0 to 198 points. Higher scores reflect greater emotional problems.
Change in behaviors as measured by the Caregiver-Teacher Report Form (C-TRF) | Baseline, 12 weeks
  The C-TRF is a 99-item, three-point Likert-type scale to assess internalizing behaviors, externalizing behaviors, attending behaviors, and aggressive in preschool-aged children. Teachers will complete the CBCL/1.5-5 pre- and post-intervention. Scores range from 0 to 198 points. Higher scores reflect greater emotional problems.

SECONDARY OUTCOMES:
Change in emotion regulation state as self-reported using the Self Assessment Manikin (SAM) | Pre-session, 20-minute post-session
  The SAM is a nonverbal, picture-based, 5-point Likert-type measure of a child's self-reported levels of pleasure (i.e., valence) and arousal (i.e., energy level). Children will complete the SAM at the beginning and end of every intervention session. Scores range from 1 to 5. Higher scores reflect greater happiness and more energy.
Change in emotion regulation state as observed using the Goal Attainment Scale (GAS) | Pre-session, 20-minute post-session
  The GAS is a way to measure individualized clinical progress on a predetermined goal, i.e. preschooler emotion regulation state. The interventionist will complete the GAS at the beginning and end of every intervention session. Scores range from negative 2 to positive 2. Higher scores reflect greater emotion regulation.
Percentage of study measures completed | 12 weeks
  Will be measured by adding the number of measures completed divided by total number of measured administered.
Percentage of child attendance | 12 weeks
  Will be measured by adding the number of study sessions completed divided by total number of study sessions.
Percentage of intervention components completed by interventionist | 12 weeks
  Measured by using a self-developed Quality Assurance (QA) checklist that tallies the number of intervention components completed. Scores will range from 0 to 100 percent, with a higher score indicating greater interventionist fidelity.

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Sena Moore, PhD, Principal Investigator — University of Miami
Locations (1):
- St. Albans Child Enrichment Center Coconut Grove, Coconut Grove, Florida, United States

IPD SHARING:
Plan to Share IPD: No